# Intestinal Microbiota Transplantation for Nonalcoholic Fatty Liver Disease (NAFLD)

Date:2017.5

# **Informed Consent Form**

#### Respected volunteer:

We are honored to invite you to take part in the research: Efficacy, Safety of Intestinal Microbiota Transplantation for Nonalcoholic Fatty Liver Disease. This study will be carried out at the Zhongshan Hospital Xiamen University. We plan to recruit 30 volunteers for. This study has been examined and approved by the ethics committee of the Medical School of Xiamen University.

The part of this article contains the rules and regulations, and in order to protect the rights and interests of the patients participating in the study. This article has been reviewed and agreed by the ethics committee.

# Why should we carry out this study?

Background:

There are trillions of microorganisms in the human intestine collectively called intestinal microbiota, which plays a crucial role in maintaining normal physiological function and intestinal immune function. Following the rising morbidity of obesity, the worldwide prevalence of nonalcoholic fatty liver disease (NAFLD) has increased and become a serious health and social problem. Intestinal microbiota may affect NAFLD through several impacts: a) increased energy harvesting and fat storage; b) impaired intestinal barrier function and consequent endotoxemia; c) systemic inflammation; d) altered choline and bile acid metabolism; e) endogenous alcohol production. Studies have indicated restore the homeostasis of intestinal microenvironment microbiota may provide the keys to new therapies for NAFLD. Intestinal microbiota transplantation is an effective way to reconstruction of the microecology of intestine which has been included in the American Medical Guide to treat Clostridium difficile infection.

Research purposes:

To investigate the efficacy and safety of intestinal microbiota transplantation for NAFLD. . Research area:

18-65 years old, corresponding to diagnosis standards of NAFLD, BMI ≥ 24.

### How does the study going on?

We plan to make the microorganisms from the fecal of the health into intestinal bacteria suspension through an intelligent processing system, and transplant it into the intestine of patients. All the patients will continue original antiviral therapy.

# What should I do in the study?

Before you participate in the study, a specialist will analyse your medical history to assess whether you are suitable for this study. If you are suitable for the study, you could sign the informed consent form and participate in the study or reject to participate in the study.

#### Do I have any other treatment options?

There is no drug treatment regimen for the treatment of NAFLD, the improvement of lifestyle such as diet and exercise is the only proven effective method in NAFLD management. You can choose:

- Do not participate in this study and continue the routine treatment, such as diet and exercise.
- Participate in other studies.
- Reject any treatment.

Please inform your doctor about your decision.

# How will this study affect my life?

We will assess your disease status. If you are suitable for the study, we will treat you with intestinal microbiota transplantation and follow up for 6 months On the basis of your informed consent form. Follow up may be inconvenient for your life. If you have any questions about the study, please consult the doctor.

#### What are the risks and adverse effects of participating in this study?

You may have an adverse effect during the study. We will monitor any adverse effects of all patients in the study. Intestinal microbiota transplantation is a relatively safe medical technique. There have been no reports of serious adverse effects so far. Short term adverse effects and complications include abdominal discomfort, abdominal distension, diarrhea, constipation, vomiting, short term fever, enteric bacterial infection, perforation and bleeding caused by endoscopic operation. We will recruit volunteers strictly according to the inclusion criteria,

monitor and deal with adverse effects that may occur. The endoscopic operation will be completed by physician with rich experience of endoscopic operation. The long-term risk include: change of the body that may caused by intestinal microbiota change like obesity, diabetes, cancer and even personality changes, etc. In order to avoid these long-term risks, we will inform the patients in detail the risks and screen the donor strictly to ensure your safety to the greatest extent. Although we have taken the preventive measures mentioned above, there is still a possibility of adverse effects even serious consequences (including death) due to the complexity of medicine, individual differences.

Therefore, we have undergone the study after examination and approval of the ethics committee and will get your informed consent form before it began. We will try our best to minimize the risk of the study as far as possible.

#### What is the reward for participating in this study?

We will exempt you from the cost of donor recruitment, acquisition of intestinal microbiota about 3000 yuan/case.

#### Is the my personal information confidential?

Your medical records will be kept in the hospital. The researchers, the research authorities, and the ethics committee will be allowed to look up the your medical records. Any public report about the results of this study will not disclose your individual identity. We will make every effort to protect the privacy of the your personal medical information within the scope of the law. Your personal and medical information will be kept confidential and kept in a safe and reliable place. You can consult the personal information, and if necessary, the information can be modified any time. When you sign this informed consent form, you agree that you agree that personal and medical information is used in the situation described above.

You sign this informed consent form only when you agree your personal and medical information will be used described above.

# Do I have to take part in the study?

It is voluntary to participate in this study. You can refuse to participate in the study or quit research without any reason anytime. The decision will not affect your future treatment. If you decide to withdraw from this study, please notify the doctor in advance. In order to ensure your safety, you may be asked to carry out related inspections, which is beneficial to the protection of

your health.

# The researchers declared:

| I confirm that the volunteer has been well informed of the details of this study, especially | |
|---|---|
| the risks and benefits that may arise from this s | tudy. f you have any questions related to this |
| project, welcome to call us anytime, and the phone | e number is +86-0592-22590151. |
| Signature of the research: | |
| The volunteers agreed to declare that: | |
| I have read the introduction of this study me | ntioned above, and I have a full understanding |
| of the risks and benefits that may arise from this st | cudy. I voluntarily participate in this clinical. |
| I agree□do not agree□ with that my medical i | records and pathological specimen in this study |
| will be used for other study. | |
| Signature of the subject: | Date: |
| Or signature of the legal representative (if there is) | : |
| Date: | |